CLINICAL TRIAL: NCT05325125
Title: Evaluating the Sequelae of Pulmonary Tuberculosis in Gambian Children
Brief Title: Childhood TB Sequel
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 22613
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children who have completed treatment for Tuberculosis: Children 19 years and below who had drug-sensitive pulmonary tuberculosis, either bacteriologically confirmed or not and who have completed treatment within the preceding 6 weeks before enrolment

SUMMARY:
This study aims to describe the long-term adverse outcomes associated with PTB in children, to describe the evolution of these sequelae, and to determine the epidemiological risk factors associated with these sequelae. The investigators will conduct a prospective cohort study. Children who have completed treatment for PTB will be enrolled. The study visit will be performed in the study clinic, where clinical assessment, spirometry and radiography will be performed. The planned duration of the study is 36 months. Participant enrolment is estimated to begin in March 2022. The estimated date of the last participant enrolled is December 2022.

DETAILED DESCRIPTION:
In the past, treatment success in TB has been defined as the eradication of active infection while preventing resistance. However, this definition of TB treatment outcome, which is based on clinical improvement and microbiological cure, is insufficient as it does not consider long-term outcomes such as loss of pulmonary function, which is medically relevant and possibly more frequent than we currently know.

With the introduction of effective treatment for PTB, the international TB community has focused more on diagnostics and therapeutics to improve disease survival. However, unlike most respiratory infections, TB tends to leave the individuals' lungs permanently destroyed or damaged. Pulmonary TB thereby transitions from a treatable communicable disease into a chronic, non-communicable disease across the life course after apparently successful treatment.

Although PTB accounts for at least 80% of the 1.2 million TB cases that occur in children, there is currently no published data about adverse health consequences and long-term impact of PTB, including changes in lung function, in children and adolescents who have completed TB treatment. However, long-term impairment in pulmonary function has been documented in more than half of the adult PTB survivors despite achieving a microbiological cure. Studies have also demonstrated that bacterial pneumonia in childhood significantly impairs the long-term function of the lungs, independent of what it was at baseline. Despite this, little is known about the changes in the pulmonary function of children after TB treatment completion, especially in low- and middle-income countries (LMIC) where the disease burden is high.

The Childhood TB Sequel study hypothesises that early childhood PTB is likely to negatively impact an individual's attained lung function and hasten the rate of decline in adulthood. While this probable impact may be subclinical in childhood, detailed prospective paediatric data are urgently needed to establish the burden of post-TB lung disease (PTLD) in children using lung function measurements regardless of symptoms and social determinants for lung health.

This study seeks to determine whether, among Gambian children and adolescents aged 19 years and below, PTB is associated with a reduction in pulmonary function measured by spirometry and an increase in the incidence of all-cause mortality. This study will include adolescents aged 15 to 19 years old who have a considerably high incidence of TB and are often neglected in childhood TB research.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19 years and below
* Reside in the Greater Banjul Area
* Were diagnosed with either confirmed or unconfirmed PTB
* Have completed treatment with an outcome of 'cured' or 'treatment completed' according to the Gambia NLTP guideline
* Parent/caregiver willing to provide written informed consent, as well as assent for the children

Exclusion Criteria:

* Relocate from the study area during the follow-up period. If they are reachable by telephone, they will be excluded from study visits in the clinic but will continue to be followed up via telephone calls
* Develop tuberculosis disease during the follow-up period

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The prevalence of TB in The Gambia is estimated to be 128 per 100,000 population, with children comprising about 8% of all notified cases annually. Over 70% of all cases of TB notified in the country reside in the GBA. The study population will comprise children and adolescents (aged 19 years and below) who are in the final month of their treatment for PTB. They will be identified for possible inclusion in the study at any of the Gambia National Leprosy and Tuberculosis Programme (NLTP) treatment clinics in the GBA. At the completion of PTB treatment, eligible children will be invited to the MRCG at LSHTM Childhood TB research clinic for formal enrolment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in self- or parent-reported respiratory symptoms | 6 months and 12 months after enrolment
  Derived from the St George's Respiratory Questionnaire and classified as 'improvement', 'no change' or 'deterioration'
Lung function measured by spirometry | 6 months and 12 months after enrolment
  The pattern of change over the 6-monthly intervals will be classified as 'improvement', 'no change' or 'deterioration' based on pre-defined minimal clinical important difference (MCID) cut-offs for the measured parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Esin Nkereuwem, MBBCh, MSc, Principal Investigator — MRCG at LSHTM
Locations (1):
- MRCG at LSHTM, Fajara, The Gambia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nkereuwem E, Agbla S, Jatta ML, Masterton U, Owolabi O, Edem VF, Kampmann B, Togun T. Childhood TB sequel: evaluating respiratory function after treatment for pulmonary tuberculosis in a prospective cohort of Gambian children - a study protocol. BMC Pulm Med. 2023 Oct 12;23(1):387. doi: 10.1186/s12890-023-02659-2. PMID 37828470